CLINICAL TRIAL: NCT00117728
Title: Clinical Relevance of Nevirapine Resistance
Brief Title: Pediatric Nevirapine Resistance Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Columbia University (Other); University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01HD047177 (NIH)
Record Dates: First submitted 2005-07-06; First posted 2005-07-08 (Estimated); Last update posted 2007-06-29 (Estimated); Status verified 2006-01

CONDITIONS: AIDS; HIV Infections
Keywords: Non-nucleoside reverse transcriptase inhibitor; Drug Resistance; HIV Seronegativity; Treatment Naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Nevirapine

INTERVENTIONS:
Drug: nevirapine

SUMMARY:
This study is designed to test if a sequential protease-inhibitor (PI) - / nevirapine (NVP) -based regimen is effective for the treatment of HIV-infected children when previous NVP exposure has occurred as part of programs to prevent mother-to-child transmission (pMTCT).

DETAILED DESCRIPTION:
The wide use of NVP in pMTCT-prophylaxis may result in resistance to NNRTI and concomitantly limits the use of these drugs for the treatment of HIV-infected children. To avoid restricting treatment options for children, it is desirable to preserve NVP for both pMTCT and first line treatment. This study will therefore test whether resistance-caused treatment failures of HIV-infected and previously NVP-exposed children can be avoided if the NVP treatment is preceded by an initial PI-based regimen.

Comparison: HIV-infected children less than 24 months of age, exposed to any pMTCT regimen that included NVP and who achieve and maintain viral suppression for at least 3 months with a PI-based regimen will be randomized to one of the two groups: (1) to continue on PI-containing regimen or (2) to be switched off the PI-containing regimen onto the NVP-containing regimen. The study outcome will be proportions in the two groups who have complete virologic suppression at 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* NVP-exposure as part of pMTCT-prophylaxis around delivery
* HIV-positive
* Eligible for treatment
* Plans to stay in the area for the next 6 months

Exclusion Criteria:

* Already on anti-retroviral treatment
* History of toxicity to perinatal NVP
* Grade 3 or greater elevation of liver function tests
* Being treated for a severe acute opportunistic infection or tumor

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2005-04; Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Virologic suppression at 6 months after randomization

SECONDARY OUTCOMES:
To compare the time to virologic failure up to 18 months post randomization
to examine the associations between detection of drug resistance mutation and virologic response to treatment
to compare the toxicity profiles and adherence in the two groups
to describe the emergence of genotypic resistance in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Louise Kuhn, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Coronation Hospital, Johannesburg, South Africa

REFERENCES:
- [Derived] Strehlau R, Kuhn L, Abrams EJ, Coovadia A. HIV-associated neurodevelopmental delay: prevalence, predictors and persistence in relation to antiretroviral therapy initiation and viral suppression. Child Care Health Dev. 2016 Nov;42(6):881-889. doi: 10.1111/cch.12399. Epub 2016 Aug 22. PMID 27546069
- [Derived] Shiau S, Kuhn L, Strehlau R, Martens L, McIlleron H, Meredith S, Wiesner L, Coovadia A, Abrams EJ, Arpadi SM. Sex differences in responses to antiretroviral treatment in South African HIV-infected children on ritonavir-boosted lopinavir- and nevirapine-based treatment. BMC Pediatr. 2014 Feb 12;14:39. doi: 10.1186/1471-2431-14-39. PMID 24521425
- [Derived] Kuhn L, Coovadia A, Strehlau R, Martens L, Hu CC, Meyers T, Sherman G, Hunt G, Persaud D, Morris L, Tsai WY, Abrams EJ. Switching children previously exposed to nevirapine to nevirapine-based treatment after initial suppression with a protease-inhibitor-based regimen: long-term follow-up of a randomised, open-label trial. Lancet Infect Dis. 2012 Jul;12(7):521-30. doi: 10.1016/S1473-3099(12)70051-8. Epub 2012 Mar 16. PMID 22424722
- [Derived] Coovadia A, Abrams EJ, Stehlau R, Meyers T, Martens L, Sherman G, Hunt G, Hu CC, Tsai WY, Morris L, Kuhn L. Reuse of nevirapine in exposed HIV-infected children after protease inhibitor-based viral suppression: a randomized controlled trial. JAMA. 2010 Sep 8;304(10):1082-90. doi: 10.1001/jama.2010.1278. PMID 20823434